CLINICAL TRIAL: NCT01007045
Title: Can Emergency Physicians Safely Exclude Proximal Deep Vein Thrombosis Using Limited Compression Emergency Department Ultrasound?
Brief Title: Limited Compression Ultrasound by Emergency Physicians to Exclude Deep Vein Thrombosis
Status: Completed | Type: Observational
Sponsor: Queen's University (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Dr. Rachel Poley, Queen's University
Other Study IDs: EMED-123-09
Record Dates: First submitted 2009-11-02; First posted 2009-11-03 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-06

CONDITIONS: Deep Vein Thrombosis
Keywords: deep vein thrombosis; venous thromboembolic disorders; diagnostic ultrasound
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Clinically "likely": Subjects deemed clinically likely to have DVT based on modified Well's criteria
- Clinically "unlikely": Subjects deemed clinically unlikely to have DVT based on modified Well's criteria

SUMMARY:
Deep vein thrombosis is a common condition seen in the Emergency Department. Standard of care for diagnosis of DVT includes a combination of a clinical pre-test probability rule known as Well's criteria, D-dimer blood testing, and Radiology department ultrasound.

The purpose of this study is to determine whether Emergency Physicians can safely rule out deep vein thrombosis using Well's criteria and D-dimer blood testing combined with Emergency department bedside ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Age > 16 years
* Clinically suspected lower extremity DVT

Exclusion Criteria:

* Known chronic DVT
* Acute DVT confirmed by prior formal imaging
* Inability to assess common femoral or popliteal area (due to cast, above knee amputation, etc.)
* Anticoagulation >48 hours prior to imaging (formal or LCU)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: emergency patients suspected of deep vein thrombosis
Sampling Method: Non-Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
First co-primary outcome: sensitivity/specificity of LC U/S vs D-dimer in clinically "unlikely" DVT patients. | 3 days
Second co-primary outcome: sensitivity/specificity of LC U/S plus D-dimer vs formal ultrasound in clinically "likely" DVT patients. | 3 days

SECONDARY OUTCOMES:
interobserver reliability of modified Well's criteria | 3 days
learning curve for LC U/S by emergency physicians and residents | 365 days
difference in diagnostic time interval for patients grouped by pre-test probability | 3 days
number of return visits for formal ultrasound imaging | 3 days
number of patients receiving empirical anticoagulation while formal ultrasound imaging is pending | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Poley, MD, Principal Investigator — Queen's University
Locations (2):
- Canada (2):
  - Kingston General Hospital, Kingston, Ontario
  - Hotel Dieu Hospital, Kingston, Ontario

REFERENCES:
- [Derived] Poley RA, Newbigging JL, Sivilotti ML. Estimated effect of an integrated approach to suspected deep venous thrombosis using limited-compression ultrasound. Acad Emerg Med. 2014 Sep;21(9):971-80. doi: 10.1111/acem.12459. PMID 25269577